CLINICAL TRIAL: NCT02498405
Title: Smartphone Twelve Lead Electrocardiogram Utility In ST-Elevation Myocardial Infarction (ST LEUIS Study)
Brief Title: Smartphone Twelve Lead Electrocardiogram Utility In ST-Elevation Myocardial Infarction
Acronym: ST LEUIS
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1040562
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to determine if the Smartphone electrocardiogram (ECG) is an acceptable replacement for a standard ECG in the identification of ST Elevation Myocardial Infarction (STEMI).

Toward this objective, this study involves the following:

* Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting with chest pain in which the STEMI protocol was activated.
* Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting to the Emergency Department for evaluation of chest pain, not necessarily presenting with STEMI.
* Reading of ECGs (standard 12-lead and iPhone) by three independent cardiologists, who are blinded to the initial clinical ECG readings, the type of ECG equipment used, and the patient's clinical information.
* Assess the operational feasibility of using the Smartphone to obtain "12-lead equivalent" ECG recordings in patients suspected to have STEMI, and
* Determine the possibility of pooling the data obtained from this study with data from other institutions conducting identical studies, and developing a future IRB-approved protocol and statistical analysis plan to compare the sensitivity, specificity, positive predictive value and the negative predictive power of the iPhone ECG, using a paired standard 12-lead ECG as the gold standard.

There will be no therapeutic interventions. A single research-related procedure will be required, i.e. an iPhone ECG. Effort will be made to ensure that the performance of this procedure will not delay any treatment and/or diagnostic procedures that are part of usual or specialized care that the patient requires. Effort will be made to enroll 1 STEMI patient for every 2 non-STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures (patient or legally acceptable representative).
* Symptoms of chest pain upon presentation at the Intermountain Medical Center Emergency Department.

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally-acceptable representative to provide written informed consent for any reason.
* Other conditions that in the opinion of the Principal Investigator or Co-Investigator(s) may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients, >18 years old, who are seen for chest pain, and/or patients for whom the STEMI protocol has been activated, will be screened for this study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis differences | 1 day
  Determine the number of agreements in diagnoses (STEMI vs. non-STEMI) between the standard 12-lead ECG and the iPhone "12-lead equivalent" ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States